CLINICAL TRIAL: NCT03626597
Title: Community-based Provision of Urine Pregnancy Tests as Linkage to Reproductive Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Moi University (Other)
Responsible Party: Principal Investigator, Caitlin Bernard, Assistant Professor, Obstetrics & Gynecology, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0003029
Record Dates: First submitted 2018-07-29; First posted 2018-08-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Prenatal Care Late; Contraceptive Usage; Pregnancy Complication
MeSH Terms: conditions — Contraception Behavior; Pregnancy Complications | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Parallel, non-blinded, patient preference model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHV-provided post-test counseling & referral (Active Comparator): The CHV will provide the woman with the urine pregnancy test and collect baseline information. If the woman desires enrollment in Arm 1 (CHV-provided post-test counseling and referral), the CHV will provide all post-test counseling and referral based on training provided. This may occur at the time of enrollment or at a later time, as preferred by the woman.
  Interventions: Diagnostic Test: Urine Pregnancy Test; Behavioral: CHV-based post-test counseling & referral
- Phone-based post-test counseling & referral (Active Comparator): The CHV will provide the woman with the urine pregnancy test and collect baseline information. If the woman desires enrollment in Arm 2 (phone-based post-test counseling and referral), the CHV will provide the woman with a phone number which she may call or short message service (SMS) to receive post-test counseling and referral. If the study team does not receive a call or SMS from the woman within one week, our research assistant will phone and/or SMS the participant to provide phone-based post-test counseling and referral.
  Interventions: Diagnostic Test: Urine Pregnancy Test; Behavioral: Phone-based post-test counseling & referral

INTERVENTIONS:
Diagnostic Test: Urine Pregnancy Test — CHV will provide all participants with in-person urine pregnancy tests (UPTs)
Behavioral: CHV-based post-test counseling & referral — CHVs will provide in-person post-test counseling & referral to care
  Arms: CHV-provided post-test counseling & referral
Behavioral: Phone-based post-test counseling & referral — Participants will call/SMS or be called/SMSed for phone-based counseling & referral to care
  Arms: Phone-based post-test counseling & referral

SUMMARY:
Kenyan families experience persistently high rates of maternal and neonatal mortality, which disproportionately affects women with low income and education and those who live far from health services. Key proven interventions include prevention of pregnancy and birth spacing, early entry to antenatal care, and facility delivery. However, creative, cost-effective interventions are urgently needed to link particularly vulnerable populations with these important health services. Previous research has shown that equipping community health volunteers (CHVs) with a tool as simple as a urine pregnancy test and training to provide post-test counseling is effective in improving linkages to antenatal care and family planning services. The invesitgators' proposal includes a multi-phase process to collect qualitative data through a needs assessment (Phase 1), use community input to develop (Phase 2) and implement a pilot intervention study (Phase 3) assessing the ability of CHV-based provision of urine pregnancy tests with CHV-provided and phone-based post-test counseling to link women with antenatal care and family planning services, and collect qualitative program evaluation data (Phase 4). This will provide much-needed information for how to effectively utilize and strengthen CHVs as part of a sustainable reproductive health care delivery system to improve maternal and neonatal mortality. The broad objectives are to determine whether the use of community-based provision of urine pregnancy tests with post-test counseling and referral to care is acceptable to community health volunteers (CHVs) and participants and to determine which method of post-test counseling and referral to care, CHV-provided or phone-based, is more acceptable and more effective. Participant outcomes, including the primary outcome of utilization of ANC or family planning care, will be measured by telephone questionnaires one to three months post-enrollment. CHV outcomes will be determined by telephone questionnaires as well as review of CHV log books.

DETAILED DESCRIPTION:
Kenyan families experience persistently high rates of maternal and neonatal morbidity and mortality, which disproportionately affects women with low educational attainment and income and those who live far from health services. Key proven interventions include prevention of pregnancy and birth spacing, early entry to antenatal care, and facility delivery. However, creative, cost-effective interventions are urgently needed to link particularly vulnerable populations with these important health services. Previous research has shown that equipping community health volunteers with a tool as simple as a urine pregnancy test and training to provide post-test counseling is effective in improving linkages to antenatal care and family planning services. The investigators' proposal includes a multi-phase process to collect qualitative data through a needs assessment, use community input to develop and implement a pilot study assessing the ability of CHV-based provision of urine pregnancy tests with CHV-provided and phone-based post-test counseling to link women with antenatal care and family planning services, and collect qualitative program evaluation data. This will provide much-needed information for how to effectively utilize and strengthen CHVs as part of a sustainable reproductive health care delivery system to improve maternal and neonatal mortality.

Expected outcomes include important qualitative data regarding the needs and preferences of women and CHVs to improve reproductive health services. Additionally, the investigators will perform a quantitative comparison of CHV-provided and phone-based post-test counseling to inform further research projects and CHV services. The investigators will plan to publish this clinical research in international peer-reviewed journals and to host community events to share the results of the study. The investigators anticipate that the outcomes from this pilot research will allow them to apply for research funding for expansion of this intervention throughout the catchment area to evaluate its effects on key population health outcomes, including maternal and neonatal mortality.

ELIGIBILITY:
CHV participants:

Inclusion:

* Approved and designated CHV by their respective county
* Has been in their role for at least 1 year Exclusion: if they do not meet the inclusion criteria

Women participants:

Inclusion Criteria:

* Women aged 15-45, inclusive
* Desire to use a urine pregnancy test for any reason.
* Have availability of a phone.
* Agree to enrollment in the study and to be contacted for data collection
* Conversant in Kiswahili or English

Exclusion Criteria:

• Physical or mental illness that precludes study involvement

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must self-represent as female
Enrollment: 308 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Utilization of care | 1-3 months post-enrollment
  Defined as proportion of participants who self-report attendance to at least one Antenatal Care (ANC) visit for women with positive UPT or Family Planning (FP) clinic visit for women with negative UPT

SECONDARY OUTCOMES:
Participant Satisfaction with CHV-based UPT provision | 1-3 months post-enrollment
  Participant self-report of satisfaction with CHV-based UPT provision on scale of very unsatisfied to very satisfied
Participant preference for CHV-based vs phone-based post-test counseling and referral | At the time of enrollment
  Proportion of participants who choose CHV-based vs. phone-based post-test counseling and referral
Number of UPTs provided per month | Monthly, thoughout the study period (estimated 10 months)
  CHV self-report of total number of UPTs provided per month (including participants & women who declined enrollment or did not meet inclusion criteria)
CHV comfort with UPT provision and post-test counseling and referral | At the time of time of UPT provision
  CHV self-report of of comfort with UPT provision and post-test counseling and referral on a scale from not comfortable to very comfortable
Participant utilization of phone-based post-test counseling and referral | 1-3 months post-enrollment
  Proportion of participants who call/SMS and respond to call/SMS for phone-based post-test counseling and referral
Results of UPTs | 1-3 months post-enrollment
  Proportion of negative vs. positive UPT results
Gestational age at first ANC visit | 1-3 months post-enrollment
  Participant self-report of gestational age at first ANC visit for women with positive UPT who attended ANC visit (reported as mean and range)
initiation of FP and method of FP | 1-3 months post-enrollment
  Participant self-report of initiation of family planning and method of family planning initiated (reported as proportion of women with negative UPT who initiated FP and proportion initiating each method of FP)

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University/MTRH, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No